CLINICAL TRIAL: NCT01649115
Title: The Healthy Lifestyles Passport Program: a Randomized Control Trial of a Prenatal Maternal Education Program to Prevent Infant and Childhood Obesity (HLPP)
Brief Title: The Healthy Lifestyles Passport Program: a Nutrition Education Program to Prevent Childhood Obesity
Acronym: HLPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bronx-Lebanon Hospital Center Health Care System (Other)
Collaborators: UnitedHealthcare Foundation (Unknown)
Responsible Party: Principal Investigator, Mamta Reddy, MD, Director, Pediatric Asthma Center; Chief, Allergy/Immunology, Bronx-Lebanon Hospital Center Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HLPP 2012
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Childhood Obesity
Keywords: obesity; overweight; childhood obesity; prevention; Z score; weight for length; WFL; body mass index; BMI; prenatal; maternal; nutrition education; health education; health literacy; health numeracy; passport; healthy lifestyles; growth; growth chart
MeSH Terms: conditions — Pediatric Obesity; Obesity; Overweight; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The Usual Care arm, will not be receiving the interactive nutrition education. They will be meeting with the Registered Dietitian twice in person after the participants are randomized in each arm, and once on the phone. The first meeting, they will be receiving pamphlets and handouts, which are typically given as part of usual care. The second meeting is a post-test assessment and Newest Vital Sign Assessment Tool. The second meeting and the follow-up phone call are both the same for usual care and the Healthy Lifestyles Passport arm.
- Healthy Lifestyles Passport (Experimental): The Healthy Lifestyles Passport arm will be receiving the intervention. They will be meeting with the Registered Dietitian twice in person after the participants are randomized into each arm, and once on the phone. The first meeting, they will be receiving the Healthy Lifestyles Passport, including the interactive nutrition education. The second meeting is a post-test assessment and Newest Vital Sign Assessment Tool.
  Interventions: Other: Healthy Lifestyles Passport

INTERVENTIONS:
Other: Healthy Lifestyles Passport — The participants will be provided with the Healthy Lifestyles Passport, and with each corresponding page, there will be an activity. Each participant in the Healthy Lifestyles Passport arm will receive the same education.
  Arms: Healthy Lifestyles Passport

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Healthy Lifestyles Passport Program (HLPP) in preventing infant and childhood obesity. It is hypothesized that the participants in the intervention arm will exhibit less excessive weight-for-length gain from 4- to 6-months of age. In 2-years and 5-years, it is predicted that the participants in the intervention arm will yield lower Body Mass Index (BMI) z-scores than the participants in the control arm, who receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women during the third trimester (>28 weeks gestation) receiving care in the institution's Women's Health Center
* no medical conditions complicating their pregnancy
* must be able to communicate in English or Spanish
* be reachable by phone
* plan to be the consistent caretaker of the child at least 75% of the time
* plan to attend the institution's pediatric outpatient clinic for the child's routine healthcare

Exclusion Criteria:

* Child with any disabling or chronic illnesses
* Any existing and/or pre-existing disabling or chronic illnesses that would qualify the mother as "high risk"
* Wards of the state
* Mothers with a disabling/serious chronic illness
* Drug/alcohol use during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in child's gender-specific weight-for-length (WFL) z-score | 4-months to 6-months of the child's age
  The child's weight and length will be extracted from the medical record at the child's 4-month and 6-month old office visit and the weight-for-length z-scores will be calculated. The difference between each arm's z-score will be compared.

SECONDARY OUTCOMES:
Child's Body Mass Index (BMI) | At 2-years and 5-years of the child's age.
  At 2-years and 5-years of age, the child's height and weight will be extracted from the medical record and BMI will be calculated. Each arm's BMI z-score will then be compared.
Mother's Knowledge, Skill, Attitude and Behavior. | Baseline, day after the intervention and two months after the baby is born.
  At baseline, all participants will answer a battery of questionnaires, including a pre-test and the "Newest Vital Sign" assessment tool. The day after the intervention, a post-test will be administered over the phone to the participants in both arms. Two months after the baby is born the same post-test and the "Newest Vital Sign" assessment tool will be administered in person.

OTHER OUTCOMES:
Change in child's gender-specific weight-for-length (WFL) z-score | 0-months to 2-months of the child's age
  The child's weight and length will be extracted from the medical record at the child's 0-month and 2-month old office visit and the weight-for-length z-scores will be calculated. The difference between each arm's z-score will be compared.
Change in child's gender-specific weight-for-length (WFL) z-score | 2-months to 4-months of the child's age
  The child's weight and length will be extracted from the medical record at the child's 2-month and 4-month old office visit and the weight-for-length z-scores will be calculated. The difference between each arm's z-score will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Reddy, MD, Principal Investigator — Bronx-Lebanon Hospital Center
Locations (1):
- Bronx-Lebanon Hospital Center, The Bronx, New York, United States